CLINICAL TRIAL: NCT02527824
Title: Phase II Study of S-1 in Combination With Oxaliplatin and Irinotecan in Patients With Advanced, Recurrent or Metastatic Biliary Tract Cancer
Brief Title: Study of Oxaliplatin, Irinotecan, and S-1 in Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hallym University Medical Center (Other)
Collaborators: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMC-HO-GI-1501
Record Dates: First submitted 2015-08-14; First posted 2015-08-19 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Biliary Tract Neoplasm
Keywords: biliary tract neoplasm; oxaliplatin; irinotecan; S-1
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Oxaliplatin; Irinotecan; S 1 (combination); gimeracil; Oxonic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxaliplatin, Irinotecan, S-1(OIS) (Experimental): intervention with triple combination chemotherapy with oxaliplatin, irinotecan, and S-1 Treatment will be delivered as a 2-week cycle.
  1. Oxaliplatin 65 mg/m2 iv on day 1
  2. Irinotecan 135 mg/m2 iv on day 1
  3. S-1 80 mg/m2/day on day 1-7
  Interventions: Drug: Oxaliplatin, Irinotecan, S-1

INTERVENTIONS:
Drug: Oxaliplatin, Irinotecan, S-1 — Treatment will be delivered every 2 weeks
  1. Oxaliplatin 65 mg/m2 iv on day 1
  2. Irinotecan 135 mg/m2 iv on day 1
  3. S-1 80 mg/m2/day on day1-7
  Other Names: Liplatin, Inotecan, TS-1(tegafur, gimeracil, oteracil)

SUMMARY:
This study will conduct a phase II study of triple combination with oxaliplatin, irinotecan, and S-1 as the first-line chemotherapy in patients with advanced biliary tract cancer.

DETAILED DESCRIPTION:
It is widely accepted that the efficacy of chemotherapy for patients with inoperable, advanced, and metastatic biliary tract cancer is better than that compared to best supportive care. In general, gemcitabine based combination chemotherapies are considered as the first line treatment for patients with advanced biliary tract cancer, but these have some limitations of inconvenience of administration and unsatisfactory efficacy.

S-1 monotherapy and combination with oxaliplatin have shown the objective response rate of 21-35% and 24.5%, respectively, and irinotecan combined with oxaliplatin has shown the response rate of 18-20.5% in patients with advanced metastatic biliary tract cancer. So the investigators had conducted the phase I study of three drugs (oxaliplatin, irinotecan, and S-1) with modification of dosage and schedule and will conduct a phase II study with recommended dose of triple chemotherapy from this phase I study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed advanced, recurrent or metastatic adenocarcinoma of biliary tract system (stage IV by primary tumor, regional nodes, metastasis(TNM) staging system)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* More than 3 months expected life span
* Measurable lesion by RECIST criteria version 1.1
* Palliative chemotherapy naive
* Adequate organ functions
* Participants must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital

Exclusion Criteria:

* Any prior 2 years or concurrent malignancy other than non-melanoma skin cancer, in situ cancer of uterine cervix, or papillary or follicular thyroid cancer.
* Participants who had received radiation therapy for target lesions 4 weeks before study enrollment
* Participants who had received major surgery 4 weeks before study enrollment
* Participants with active infection, severe heart disease, uncontrollable hypertension or diabetes mellitus, myocardial infarction during the preceding 12 months, pregnancy, or breast feeding
* Participants with central nervous system(CNS) metastases
* Participants with peripheral sensory neuropathies with impaired functional activities
* Participants with gastrointestinal obstruction or bleeding inducing mal-absorption of oral chemotherapeutic agents.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-08 (Actual); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 1.5 year
  Tumor response will be classified on the basis of the response evaluation criteria in solid tumors (RECIST) guidelines version 1.1

SECONDARY OUTCOMES:
progression free survival | 1.5 year
  The progression-free survival (PFS) will be measured from the start of study treatment until documented tumor progression (by RECIST) or death due to any cause
overall survival | 1.5 year
  The overall survival (OS) will be estimated from the start of study treatment until participant's death and measured using the Kaplan-Meier method
toxicity profiles - the number of participants and grade of intensity of treatment related adverse events | 1.5 year
  adverse events will be graded using the NCI common terminology criteria for adverse events (NCTCAE) v 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Dae Young Zang, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym university medical center, Anyang, Gyunggi, South Korea

IPD SHARING:
Plan to Share IPD: Undecided